CLINICAL TRIAL: NCT01971580
Title: The Effects of Ambrisentan on Exercise Capacity in Fontan Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, Ari Cedars, Assistant Professor of Medicine, Washington University School of Medicine
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IN-US-300-D076
Record Dates: First submitted 2013-10-23; First posted 2013-10-29 (Estimated); Results first posted 2018-05-07 (Actual); Last update posted 2018-05-07 (Actual); Status verified 2018-05

CONDITIONS: Single Ventricle Fontan Palliation
MeSH Terms: interventions — ambrisentan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ambrisentan first, Placebo second (Other): These patients will be randomized to have ambrisentan during the first study period, and placebo during the second study period.
  Interventions: Drug: Ambrisentan
- Placebo first, Ambrisentan second (Other): These patients will be randomized to have placebo during the first study period, and ambrisentan during the second study period.
  Interventions: Drug: Ambrisentan

INTERVENTIONS:
Drug: Ambrisentan
  Other Names: Letaris

SUMMARY:
Hypothesis:

Patients with a Fontan type palliation are limited by preload, or the rate at which blood returns to the heart after passively traversing the pulmonary capillary bed. By decreasing pulmonary vascular resistance using an endothelin receptor antagonist, both ventricular filling pressures and volumes will increase with a simultaneous decrease in systemic impedance to flow and decrease in central venous pressures, leading to an improved capacity to increase cardiac output, and thereby an improvement in patient functional status.

Patients who are candidates for the study will be randomized to a double-blind single crossover study. Therapy with either ambrisentan or placebo will be continued for 12 weeks, with a 2 week washout period between treatment periods. Subjects will be subjected to a VO2 max test to evaluate exercise capacity at enrolment, and on the last day of each treatment period. As a component of the VO2 max testing the patient's VE, VCO2, VE/VCO2 slope, ventilatory anaerobic threshold (VAT), peak work, efficiency, and other physiologic parameters as typically obtained from cardiopulmonary testing will be assessed. In addition, each patient will be asked to complete an SF-36 quality of life questionnaire at enrollment, and on the last day of each study period.

ELIGIBILITY:
Inclusion Criteria:

1. Patients over 18 years of age followed at the Center for Adults with Congenital Heart Disease at Washington University School of Medicine or at Saint Louis Childrens Hospital who have had a Fontan-type of palliation with single ventricular physiology.
2. Patients must not within the last year have been treated with an endothelin receptor antagonist, phosphodiesterase 5 antagonist, or prostacyclin analogue.
3. Female patients must not be pregnant, and during the study period must be using effective contraception (including barrier method with spermicide, intrauterine device, implanon, oral contraceptives) if fertile.
4. In the physicians opinion patients must be able to complete a VO2 max test to achieve an RER of >1.0
5. In the physicians opinion patients must be socially and intellectually able to adhere to the treatment regimen and follow-up
6. Patients must be intellectually able to reliably complete an SF-36 questionnaire on quality of life.
7. Patients must be clinically stable for at least 3 months prior to enrolment.
8. Patients must not have had surgery within 6 months prior to enrolment, and have no planned surgery for the study period.
9. Patients must provide informed consent.

   -

Exclusion Criteria:

1. Patients under 18 years of age.
2. Patients who are pregnant, nursing, or who in the physician's opinion are likely to become pregnant.
3. Patients who are clinically unstable.
4. Patients who have previously been treated with either an endothelin receptor antagonist and stopped due to adverse side effects.
5. Patients with an AST or ALT of >3 x normal.
6. Patients having any known contraindication to the initiation of ambrisentan.
7. Patients with a calculated creatinine clearance of <60ml/min
8. Patients with a serum hemoglobin concentration of <10mg/dl
9. Patients with a poorly controlled cardiac arrhythmia
10. Patients who are unable to provide independent informed consent.

    -

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2012-08; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from Washington University School of Medicine Adult Congenital Heart Disease clinic between 10/2012 and 11/2014
Groups:
- Ambrisentan First, Placebo Second: These patients will be randomized to have ambrisentan during the first study period, and placebo during the second study period.
  Ambrisentan
- Placebo First, Ambrisentan Second: These patients will be randomized to have placebo during the first study period, and ambrisentan during the second study period.
  Ambrisentan
Period: Overall Study
Arm/Group | Ambrisentan First, Placebo Second | Placebo First, Ambrisentan Second
Started | 14 | 14
Completed | 10 | 9
Not Completed | 4 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ambrisentan First, Placebo Second | Placebo First, Ambrisentan Second | Total
Number analyzed (Participants) | 14 | 14 | 28
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 14 | 14 | 28
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 4 | 11
  Male | 7 | 10 | 17

OUTCOME MEASURES:

1. Primary Outcome: Change in VO2 Max
Time Frame: Baseline compared to 12 weeks therapy with either ambrisentan or placebo
Population: In this crossover study, all patients received both ambrisentan and placebo. Data was analyzed comparing baseline measures to those after the period on ambrisentan and baseline measures to those after the period on placebo.
Measure: Mean (95% Confidence Interval); unit: Change in ml/kg min
Groups:
- On Ambrisentan Therapy: After Ambrisentan compared to baseline
- On Placebo: After Placebo compared to baseline
Arm/Group | On Ambrisentan Therapy | On Placebo
Number analyzed (Participants) | 19 | 19
Change in ml/kg min | 1.33 [-0.92 to 3.57] | 0.745 [-2.06 to 2.42]

2. Secondary Outcome: Quality of Life
Description: Change in Rand 36-item Short Form (SF-36) physical function score (0-100). On the Rand SF-36 questionnaire, a score closer to 100 (higher) suggests lesser disability, while a score closer to 0 (lower) suggests more disability.
Time Frame: 12 weeks
Population: In this crossover study, all patients received both therapies. Analysis was performed comparing baseline to after indicated therapy
Measure: Mean (95% Confidence Interval); unit: Change in score from baseline
Groups:
- On Ambrisentan Therapy: Baseline compared to after period of ambrisentan therapy
- On Placebo: Baseline compared to after placebo therapy
Arm/Group | On Ambrisentan Therapy | On Placebo
Number analyzed (Participants) | 19 | 19
Change in score from baseline | 3.75 [-5.78 to 13.2] | 0.195 [-9.34 to 9.73]

ADVERSE EVENTS:
Time Frame: During the study period and for one month after the completion of the study protocol, an average of 30 weeks.
Groups:
- On Ambrisentan Therapy: Events that occurred while on ambrisentan therapy
- On Placebo: Events that occurred while on placebo therapy
Arm/Group | On Ambrisentan Therapy | On Placebo
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/19
Serious Adverse Events (participants affected / at risk) | 1/19 | 0/19
Other Adverse Events (participants affected / at risk) | 13/19 | 14/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | On Ambrisentan Therapy (N=19) | On Placebo (N=19)
Gastroenteritis and acidosis (Gastrointestinal disorders) | 1 (1) | 0 (0) — Subject developed a viral gastroenteritis not related to drug therapy which provoked drug discontinuation and hospitalization. The subject was still interested in participating and after recovering restarted the study protocol without problems.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | On Ambrisentan Therapy (N=19) | On Placebo (N=19)
Rhinitis or Pharyngitis (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 8 (8)
edema (Skin and subcutaneous tissue disorders) | 3 (3) | 2 (2)
rash (Skin and subcutaneous tissue disorders) | 2 (2) | 3 (3)
arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
cough/dyspnea (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 3 (3)
nausea (Gastrointestinal disorders) | 4 (4) | 2 (2)
chest pain (Cardiac disorders) | 0 (0) | 2 (2)
fatigue (General disorders) | 1 (1) | 1 (1)
abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
diarrhea (Gastrointestinal disorders) | 1 (1) | 2 (2)

LIMITATIONS AND CAVEATS:
Large dropout rate. Small sample size. Many individuals did not achieve the target RER during cardiopulmonary exercise testing.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No